CLINICAL TRIAL: NCT00106327
Title: Improving Functioning in Peripheral Arterial Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Mary McDermott, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 171; R01HL073351 (NIH)
Record Dates: First submitted 2005-03-22; First posted 2005-03-23 (Estimated); Last update posted 2012-07-25 (Estimated); Status verified 2012-07

CONDITIONS: Cardiovascular Diseases; Peripheral Vascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Peripheral Vascular Diseases | interventions — Exercise; Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- 1 (Experimental): 6-month supervised treadmill exercise program
  Interventions: Behavioral: Exercise
- 2 (Experimental): 6-month supervised lower extremity progressive resistance training program
  Interventions: Behavioral: Exercise
- 3 (Active Comparator): Diet/nutrition control group
  Interventions: Behavioral: Diet

INTERVENTIONS:
Behavioral: Exercise — 6 months of supervised treadmill exercise or strength training, three times per week, followed by a 6 month home-based program.
  Arms: 1; 2
Behavioral: Diet — 11 nutrition education sessions
  Arms: 3

SUMMARY:
The purpose of this study is to compare the effects of nutrition, a supervised treadmill exercise program, and supervised progressive resistance training program on peripheral arterial disease.

DETAILED DESCRIPTION:
BACKGROUND:

Previous work demonstrates that functional limitations associated with peripheral arterial disease (PAD) are diverse and include slower walking speed, poorer walking endurance, and impaired balance as compared to persons without PAD. Although treadmill-walking exercise improves treadmill performance in patients with intermittent claudication (IC), treadmill performance does not correlate well with community walking ability in older men and women. In older patient populations without PAD, resistance training improves functioning and walking endurance, but this mode of exercise has not been sufficiently studied in PAD. Furthermore, although 65% to 70% of men and women with PAD are either asymptomatic or have exertional leg symptoms other than IC, no prior studies have assessed the effects of exercise interventions in PAD patients who do not have IC.

DESIGN NARRATIVE:

The randomized, control study will determine whether a 6-month supervised treadmill exercise program and a supervised lower extremity progressive resistance training program, respectively, improve lower extremity functioning compared to a nutrition control group among 150 PAD patients with and without IC. The investigators hypothesize that participants in the treadmill walking exercise program and participants in the progressive resistance training program, respectively, will experience greater improvement in functional outcomes than participants in the nutrition control group. The primary functional outcome measures in descending order of importance are 6-minute walk distance and the summary performance score. The summary performance score is a composite measure of lower extremity functioning (usual walking speed, standing balance, and time required for five repeated chair rises) measured on a 0-12 scale that predicts future risk of nursing home placement, mobility loss, and mortality. The study will also identify mechanisms by which the exercise interventions improve functioning in PAD. Mechanisms to be studied include changes in blood viscosity, calf blood flow, brachial artery endothelial reactivity, and inflammatory cytokine levels. By identifying the optimal exercise program for improving functioning in PAD patients with and without IC, the findings will have substantial clinical and public health implications for millions of patients with PAD.

ELIGIBILITY:
Inclusion Criteria:

* 150 peripheral arterial disease patients with and without IC

Exclusion Criteria:

* Below or above-knee amputation
* Wheelchair confinement
* Inability to walk on a treadmill or inability to perform progressive resistance training
* Inability to return to the medical center three times weekly for 6 months
* Walking impairment due to a cause other than PAD
* Class II New York Heart Association (NYHA) heart failure or angina (heart failure or angina occurring at rest or with minimal exertion)
* Planned lower extremity revascularization or any other major surgery within 12 months
* Any increase in anginal symptoms during the previous 6 months or angina at rest
* Subjects with silent coronary ischemia, defined as ST segment depression greater than or equal to 1 mm during baseline exercise treadmill test without associated chest discomfort, unless they have had a normal perfusion stress test during the previous 6 months
* Subjects with left-bundle branch block or significant ST-T wave changes on their baseline ECG who do not have a perfusion stress test demonstrating absence of reversible ischemia within the previous 6 months
* Lower extremity revascularization, major orthopedic surgery, or other major surgery during the previous 3 months
* Myocardial infarction or coronary artery bypass grafting during the previous 3 months
* Major medical illnesses that may interfere with subject's ability to complete the interventions and/or follow-up testing
* Current foot ulcer
* ABI greater than 0.95
* Life expectancy less than 12 months
* Does not speak English
* Patient is currently involved in another clinical trial
* Dementia
* Poorly controlled blood pressure
* Current significant exercise, defined as exercising three times weekly for 30 minutes with sufficient exertion to produce a sweat or other exercise that is comparable to the exercise interventions offered in our protocol
* Treatment for cancer (other than non-melanoma skin cancer) during the past 12 months (including radiation therapy, chemotherapy, or surgery)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2003-09; Primary Completion 2008-07 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Six-minute walk distance | Measured at baseline and follow-up study visits
Summary performance score | Measured at baseline and follow-up study visits

CONTACTS AND LOCATIONS:
Overall Officials: Mary McDermott, MD, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

REFERENCES:
- [Derived] Hammond MM, Tian L, Zhao L, Zhang D, McDermott MM. Attendance at Supervised Exercise Sessions and Walking Outcomes in Peripheral Artery Disease: Results From 2 Randomized Clinical Trials. J Am Heart Assoc. 2022 Dec 20;11(24):e026136. doi: 10.1161/JAHA.122.026136. Epub 2022 Dec 19. PMID 36533626
- [Derived] McDermott MM, Tian L, Criqui MH, Ferrucci L, Greenland P, Guralnik JM, Kibbe MR, Li L, Sufit R, Zhao L, Polonsky TS. Perceived Versus Objective Change in Walking Ability in Peripheral Artery Disease: Results from 3 Randomized Clinical Trials of Exercise Therapy. J Am Heart Assoc. 2021 Jun 15;10(12):e017609. doi: 10.1161/JAHA.120.017609. Epub 2021 Jun 2. PMID 34075780
- [Derived] Patel K, Polonsky TS, Kibbe MR, Guralnik JM, Tian L, Ferrucci L, Criqui MH, Sufit R, Leeuwenburgh C, Zhang D, Zhao L, McDermott MM. Clinical characteristics and response to supervised exercise therapy of people with lower extremity peripheral artery disease. J Vasc Surg. 2021 Feb;73(2):608-625. doi: 10.1016/j.jvs.2020.04.498. Epub 2020 May 19. PMID 32416309
- [Derived] McDermott MM, Kibbe MR, Guralnik JM, Ferrucci L, Criqui MH, Domanchuk K, Tian L, Zhao L, Li L, Patel K, Polonsky TS. Durability of Benefits From Supervised Treadmill Exercise in People With Peripheral Artery Disease. J Am Heart Assoc. 2019 Jan 8;8(1):e009380. doi: 10.1161/JAHA.118.009380. PMID 30587066
- [Derived] McDermott MM, Ferrucci L, Guralnik JM, Dyer AR, Liu K, Pearce WH, Clark E, Liao Y, Criqui MH. The ankle-brachial index is associated with the magnitude of impaired walking endurance among men and women with peripheral arterial disease. Vasc Med. 2010 Aug;15(4):251-7. doi: 10.1177/1358863X10365181. Epub 2010 May 28. PMID 20511294
- [Derived] Payvandi L, Dyer A, McPherson D, Ades P, Stein J, Liu K, Ferrucci L, Criqui MH, Guralnik JM, Lloyd-Jones D, Kibbe MR, Liang ST, Kane B, Pearce WH, Verta M, McCarthy WJ, Schneider JR, Shroff A, McDermott MM. Physical activity during daily life and brachial artery flow-mediated dilation in peripheral arterial disease. Vasc Med. 2009 Aug;14(3):193-201. doi: 10.1177/1358863X08101018. PMID 19651668
- [Derived] McDermott MM, Ades P, Guralnik JM, Dyer A, Ferrucci L, Liu K, Nelson M, Lloyd-Jones D, Van Horn L, Garside D, Kibbe M, Domanchuk K, Stein JH, Liao Y, Tao H, Green D, Pearce WH, Schneider JR, McPherson D, Laing ST, McCarthy WJ, Shroff A, Criqui MH. Treadmill exercise and resistance training in patients with peripheral arterial disease with and without intermittent claudication: a randomized controlled trial. JAMA. 2009 Jan 14;301(2):165-74. doi: 10.1001/jama.2008.962. PMID 19141764
- [Derived] McDermott MM, Ades PA, Dyer A, Guralnik JM, Kibbe M, Criqui MH. Corridor-based functional performance measures correlate better with physical activity during daily life than treadmill measures in persons with peripheral arterial disease. J Vasc Surg. 2008 Nov;48(5):1231-7, 1237.e1. doi: 10.1016/j.jvs.2008.06.050. Epub 2008 Oct 1. PMID 18829215